CLINICAL TRIAL: NCT01157039
Title: A Phase II Trial of Glutamin to Prevent Oxaliplatin Neurotoxicity and a Pharmacokinetic Analysis of Oxaliplatin.
Brief Title: A Trial of Glutamine to Prevent Oxaliplatin Neurotoxicity and a Pharmacokinetic Analysis of Oxaliplatin
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: abandoned
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 25070
Record Dates: First submitted 2010-07-02; First posted 2010-07-05 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2011-10

CONDITIONS: Colorectal Carcinoma; Neoplasms, Colorectal; Colorectal Cancer; Colorectal Tumors; Metastasis
Keywords: glutamine; oxaliplatin; adverse effects
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Glutamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dietary Supplement (Experimental): Arm A: At cycle 2, patients will be randomized to receive for 6 days- Glutamine 30g/day during cycle 2 and glutamine 40g/day during cycle 3
  Interventions: Dietary Supplement: Glutamine
- Dietary supplement (Experimental): Arm B: At cycle 2, patients will be randomized to receive for 6 days: Glutamine 40g/day at cycle 2 and glutamine 30g/day at cycle 3.
  Interventions: Dietary Supplement: Glutamine

INTERVENTIONS:
Dietary Supplement: Glutamine — Glutamine- During the first cycle of oxaliplatin based combination therapy (mFOLFOX 6 or XELOX) no patient will receive glutamine. At cycle 2, patients will be randomized to receive for 6 days either : Glutamine 30g/day during cycle 2 and glutamine 40g/day during cycle 3 (ARM A) or glutamine 40g/day at cycle 2 and glutamine 30g/day at cycle 3 (Arm B).
  Other Names: L-glutamine

SUMMARY:
The investigators hypothesize that glutamine significantly reduces the incidence and severity of peripheral neuropathy in patients receiving oxaliplatin for metastatic colorectal cancer, decreases the need for dose reduction of oxaliplatin, and it does not impair oxaliplatin efficacy or pharmacokinetics.

DETAILED DESCRIPTION:
This is a phase II , open-label, non randomized study of oral glutamine administration to evaluate oxaliplatin pharmacokinetics, and to prevent oxaliplatin neurotoxicity in patients with metastatic colorectal cancer.

ELIGIBILITY:
Study Population: The target population is patients with metastatic colorectal adenocarcinoma who are sufficiently robust to undergo at least 3 cycles of oxaliplatin based chemotherapy (mFOLFOX or XELOX) Sampling Method: Probability Sample.

Inclusion Criteria:

* Patients must hvae metastatic colorectal cancer (stage IV)
* Patients who have been treated with FOLFIRI regimen for metastatic setting may be eligible for this trial
* Patients must be ≥ 18 years
* Patients must have an Eastern Cooperative Oncology Group (EGOC) performance status 0 to 2.
* Patients must have adequate renal function of creatinine < 1.5mg/dL and a creatinine clearance > 45mL/min; patients must have adequate hepatic function with a bilirubin < 1.5mg/dL and AST (normal range 0-14 U/L) and ALT (normal range 0-49 U/L); and patients must have adequate bone marrow function with absolute neutrophil count (ANC) ≥ 1,500/цL and platelets ≥ 100,000/цL and a hemoglobin ≥ 10g/d.
* Patients must be willing and able to comply with the study protocol for the duration of the study.
* Patients must give written informed consent prior to any study-specific screening procedures with the understanding that the patient may withdraw consent at any time without prejudice.
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment. Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation.
* The investigator is requested to advise the patient how to achieve an adequate contraception
* Life expectancy longer than 6 months

Exclusion Criteria:

* Patients who have received oxaliplatin previously
* Patients with previous of current diagnosis of peripheral sensory neuropathy
* Patients who have tested positive for HIV
* Patients with other significant medical, psychiatric disorders that, in the opinion of the investigator, will exclude the patient from the study for compliance or safety reasons.
* Patients who cannot swallow
* History of known allergy to oxaliplatin or other platinum compounds, to 5-FU, to LV, glutamine or to any ingredients in the formulations of the containers
* Participation in another clinical trial with any investigational drug within 30 days prior to study screening.
* Pernicious anemia or other megaloblastic anemia with vitamin B12 deficiency
* Patients with concomitant treatment with drugs/ingredients reported to have a potential activity to prevent PSN
* Patients who haven't successfully completed local therapy for previously treated CNS metastases and who haven't been discontinued with corticosteroid for > 4wks before starting chemotherapy. Patients with asymptomatic brain mets. who have no evidence of midline shift on CT/ MRI may be enrolled without initiation of local therapy for the CNS mets. Repeat scan must be preformed < 4wks to ensure no progression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-10; Primary Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
To evaluate potential pharmacokinetic interactions between oxaliplatin and glutamine at 30g and 40g in patients with metastatic colorectal cancer. | Post cycle 2 and cycle 3

SECONDARY OUTCOMES:
To evaluate effects of glutamine supplementation on neuropathy and diarrhea related to oxaliplatin, and on dose reductions and in patients with metastatic colorectal cancer. | Post cycle 2 to 30-day follow-up visit
To compare the toxicity profile of glutamine and FOLFOX to historical data. | Post cycle 2 to 30-day follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sawyer, MD, Study Chair — Alberta Health services